CLINICAL TRIAL: NCT05115110
Title: A Two-Part, Seamless, Multi-Center, Randomized, Placebo-Controlled, Double-Blind Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of RO7204239 in Combination With Risdiplam (RO7034067) in Patients With Spinal Muscular Atrophy
Brief Title: A Study to Investigate the Safety and Efficacy of RO7204239 in Combination With Risdiplam (RO7034067) in Participants With Spinal Muscular Atrophy
Acronym: MANATEE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN42644; 2023-506761-65-00 (Other: CTIS (EU CTR))
Record Dates: First submitted 2021-11-01; First posted 2021-11-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7204239 + Risdiplam (Experimental): Participants who have not previously been treated with risdiplam will receive risdiplam for at least 8 weeks prior to randomization into a treatment group (Part 1 only). Participants that have been treated with risdiplam for at least 8 continuous weeks immediately prior to joining the study may be immediately randomized to combination therapy, or join the study run-in period (the period between screening and randomization to a treatment group) where they will continue to receive risdiplam monotherapy until randomization.
  Participants enrolled in Part 1 will receive RO7204239 (low or high dose) + risdiplam for 24 weeks, followed by RO7204239 + risdiplam for 72 weeks.
  Participants enrolled in Part 2 will receive risdiplam for 8 weeks and then treatment with RO7204239 + risdiplam for 72 weeks.
  Once the treatment period has completed (Part 1 or Part 2), participants will have the option of treatment with RO7204239 + risdiplam for 2 additional years.
  Interventions: Drug: RO7204239; Drug: Risdiplam
- Placebo + Risdiplam (Active Comparator): Participants who have not previously been treated with risdiplam will receive risdiplam for at least 8 weeks prior to randomization into a treatment group (Part 1 only). Participants that have been treated with risdiplam for at least 8 continuous weeks immediately prior to joining the study may be immediately randomized to combination therapy, or join the study run-in period (the period between screening and randomization to a treatment group) where they will continue to receive risdiplam monotherapy until randomization.
  Participants enrolled in Part 1 will receive placebo (low or high dose-matched) + risdiplam for 24 weeks, followed by RO7204239 + risdiplam for 72 weeks.
  Participants enrolled in Part 2 will receive risdiplam for 8 weeks and then treatment with placebo + risdiplam for 72 weeks.
  Once the treatment period has completed (Part 1 or Part 2), participants will have the option of treatment with RO7204239 + risdiplam for 2 additional years.
  Interventions: Drug: Placebo; Drug: Risdiplam

INTERVENTIONS:
Drug: RO7204239 — RO7204239 will administered every 4 weeks (Q4W) by subcutaneous (SC) injection into the abdomen.
  RO7204239 will be investigated at low- and high-dose in Part 1.
  Arms: RO7204239 + Risdiplam
Drug: Placebo — Placebo will be administered Q4W by SC injection into the abdomen.
  Arms: Placebo + Risdiplam
Drug: Risdiplam — Risdiplam will be administered orally once daily (QD) for the duration of the study.
  Other Names: RO7034067; Evrysdi

SUMMARY:
Risdiplam works by helping the body produce more survival motor neuron (SMN) protein throughout the body. This means fewer motor neurons - nerve cells that pass impulses from nerves to muscles to cause movement - are lost, which may improve how well muscles work in people with SMA. RO7204239 is an investigational anti-myostatin antibody that is designed to target myostatin. Myostatin plays an important role in the regulation of skeletal muscle size by controlling growth. Inhibiting myostatin may help muscles grow in size and strength. RO7204239 in combination with risdiplam, which is designed to increase the amount of SMN protein throughout the body, has the potential to further improve motor function and clinical outcomes for people living with SMA.

This trial will study the safety and efficacy of RO7204239 in combination with risdiplam in patients with spinal muscular atrophy (SMA). The trial has two parts; Part 1 is the dose-finding part in SMA patients that are either ambulant (aged 2-10 years) or non-ambulant (aged 5-10 years) within separate cohorts, and Part 2 is the pivotal part in SMA patients aged 2-25 years that are ambulant.

ELIGIBILITY:
Inclusion Criteria:

* Age at screening: Part 1 Cohorts A (ambulant participants), B (ambulant participants), and D (non-ambulant participants): 5-10 years, inclusive; Part 1 Cohort C (ambulant participants): 2-4 years, inclusive; Part 2 (ambulant participants): 2-25 years, inclusive
* Participants who have a confirmed genetic diagnosis of 5q-autosomal recessive SMA
* Symptomatic SMA disease, as per investigator's clinical judgement
* Participants who have received previous SMA disease-modifying therapies may be included provided that: Onasemnogene abeparvovec was received at least 90 days prior to screening. Participants should be tapered off steroids prior to receiving risdiplam. In addition, participants should have normal levels of liver function tests, coagulatory parameters, platelets, and troponin-I at 90 days after administration of onasemnogene abeparvovec or at least 1 month after tapering off corticosteroids, whichever comes later; Nusinersen last dose was received at least 90 days prior to screening; Risdiplam is switched to the investigational medicinal product (IMP) provided by the site

Inclusion Criteria for Part 1 Cohorts A, B, and C and Part 2 only:

* Participants who are ambulant, where ambulant is defined as able to walk/run unassisted (i.e., without the use of assistive devices such as canes, walking sticks, crutches, walkers, person/hand-held assistance, braces, orthoses, over the malleoli insoles or any other type of support) 10 meters in ≤ 30 seconds as measures by the Timed 10-Meter Walk/Run Test [10MWRT] at screening

Inclusion Criteria for Part 1 Cohort D only:

* Participants who are able to sit, defined by: A score of 3 on Item 9 of the MFM32 (sitting without upper limb support while maintaining contact between the two hands for 5 seconds); A score of at least 2 on Item 10 of the MFM32 (while seated, leaning forward to touch a tennis ball and sitting back again, either with or without upper limb support)
* Participants who are able to raise a standardized plastic cup with a 200g weight in it to the mouth, using both hands if necessary, defined by a score of 3 on the entry item of the Revised Upper Limb Module (RULM)

Exclusion Criteria:

* Concomitant or previous participation in any investigational drug or device study within 90 days prior to screening or 5 half-lives of the drug whichever is longer, with the exception of those who have completed a risdiplam study, or participated in a nusinersen or onasemnogene abeparvovec study
* Receiving or have received previous administration of anti-myostatin therapies
* Any history of cell therapy
* Hospitalization for a pulmonary event within the last 2 months or planned hospitalization at the time of screening
* Past surgery for scoliosis or hip fixation in the 6 months preceding screening or planned within the next 9 months (Part 1) or 21 months (Part 2)
* Unstable gastrointestinal, renal, hepatic, endocrine, or cardiovascular system diseases considered to be clinically significant
* Clinically significant ECG abnormalities at screening from average of triplicate measurement, abnormal findings at echocardiography, or cardiovascular disease indicating a safety risk for participants at the time of screening
* Any major illness within 1 month before screening
* Received any multidrug and toxin extrusion (MATE1/2K) substrates within 2 weeks before screening
* Hereditary fructose intolerance
* Used any of the following medications within 90 days prior to screening: riluzole, valproic acid, hydroxyurea, sodium phenylbutyrate, butyrate derivatives, creatine, carnitine, growth hormone, anabolic steroids, probenecid, acetyl cholinesterase inhibitors, agents that could potentially increase or decrease muscle strength, and agents with known or presumed histone deacetylase (HDAC) inhibitory effect
* Clinically significant abnormalities in laboratory test results at the time of screening
* Ascertained or presumptive hypersensitivity to RO7204239 or risdiplam, or to the constituents of its formulations
* Clinically relevant history of anaphylactic reaction requiring inotropic support
* Any abnormal skin conditions, pigmentation or lesions in the area intended for SC injection (abdomen) and that would prevent visualization of potential injection site reactions to RO7204239
* Immobilization, surgical procedures, fracture, or trauma to the upper or lower limbs within 90 days prior to screening

Exclusion Criteria for Part 1 Cohorts A and B only:

* Participants with contraindications for MRI scan (including, but not restricted to, claustrophobia, pacemaker, artificial heart valves, cochlear implants, presence of foreign metal objects in heart or body, including spinal rods, intracranial vascular clips, insulin pumps, etc.), difficulties maintaining a prolonged supine position, or any other clinical history or examination finding that would pose a potential hazard in combination with MRI

Exclusion Criteria for Part 1 Cohort D only:

* Participants who are unable to adopt the correct position to endure adequate quality of DXA scan acquisition, as determined by the DXA scan technologist
* Participants who have contractures at screening that would interfere with DXA scan acquisition or functional assessments, as confirmed by the DXA scan technologist and clinical evaluator
* For participants able to take steps only: Able to walk unassisted (i.e., without the use of assistive devices such as canes, walking sticks, crutches, walkers, person/hand held assistance, braces, orthoses, over the malleoli insoles or any other type of support) 10 meters in ≤ 30 seconds as measured by the timed 10MWRT at screening
* Participants who have severe scoliosis (curvature > 40°) at screening based on the participant's most recent X-ray as performed per standard of care or scoliosis that would interfere with functional assessments, as confirmed by the clinical evaluator. An X-ray is not required if it is not clinically indicated (e.g., in participants with mild scoliosis)
* Participants who require invasive ventilation, tracheostomy, or the use of noninvasive ventilation (e.g., bilevel positive airway pressure) during the daytime

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 259 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2029-02-27 (Estimated); Study Completion 2029-02-27 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Percentage of participants with adverse events (AEs) | Up to 4.5 years
Part 1 - Incidence of relevant echocardiographic parameter z scores > 2 | Up to 4.5 years
Part 1 - Serum concentration of RO7204239 | Through Week 96
Part 1 - Time to maximum serum concentration (Cmax) of RO7204239 | Through Week 96
Part 1 - Area under the curve (AUC) of RO7204239 | Through Week 96
Part 1 - Trough concentration (Ctrough) of RO7204239 | Through Week 96
Part 1 - Plasma concentration of risdiplam | Week 21
Part 1 - Plasma concentration of risdiplam metabolite (M1) | Week 21
Part 1 - Cmax of risdiplam | Week 21
Part 1 - AUC of risdiplam | Week 21
Part 1 - Ctrough of risdiplam | Week 21
Part 1 - Incidence of anti-drug antibodies (ADAs) | Through Week 96
Part 1 - Change from baseline in serum concentration of total myostatin | Through Week 85
Part 1 - Change from baseline in serum concentration of free latent myostatin | Through Week 85
Part 1 - Change from baseline in serum concentration of mature myostatin | Through Week 85
Part 1 - Percent change from baseline in the contractile area of skeletal muscle in the dominant thigh muscles as assessed by magnetic resonance imaging (MRI) in participants aged at least 5 years | Week 24 of combination treatment
Part 1 - Percent change from baseline in the contractile area of skeletal muscle in the dominant calf muscles as assessed by MRI in participants aged at least 5 years | Week 24 of combination treatment
Part 2 - Change from baseline in Revised Hammersmith Scale (RHS) total score | Week 72 of combination treatment (study Week 80)

SECONDARY OUTCOMES:
Part 2 - Change from baseline in Motor Function Measure (MFM) Domain 1 + Domain 2 (D1 + D2) score | Week 72 of combination treatment (study Week 80)
Part 2 - Change from baseline in MFM-32 total score | Week 72 of combination treatment (study Week 80)
Part 2 - Change from baseline in time taken to rise from the floor as measured by RHS Item 25 | Week 72 of combination treatment (study Week 80)
Part 2 - Change from baseline in time taken to walk/run 10 meters as measured by RHS Item 19 | Week 72 of combination treatment (study Week 80)
Part 2 - Percent change from baseline in lean mass as assessed by full body dual energy X-ray absorptiometry (DXA) scan in participants aged at least 5 years | Week 72 of combination treatment (study Week 80)
Part 2 - Percentage of participants with adverse events (AEs) | Up to 4.5 years
Part 2 - Serum concentration of RO7204239 | Through Week 80
Part 2 - Cmax of RO7204239 | Through Week 80
Part 2 - AUC of RO7204239 | Through Week 80
Part 2 - Ctrough of RO7204239 | Through Week 80
Part 2 - Plasma concentration of risdiplam | Week 32
Part 2 - Plasma concentration of risdiplam metabolite (M1) | Week 32
Part 2 - Cmax of risdiplam | Week 32
Part 2 - AUC of risdiplam | Week 32
Part 2 - Ctrough of risdiplam | Week 32
Part 2 - Incidence of ADAs | Through Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- United States (4):
  - Nemours Children's Hospital, Orlando, Florida
  - Boston Childrens Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Neurology & Neuromuscular Care Center, Denton, Texas
- Sydney Children's Hospital, Randwick, New South Wales, Australia
- Belgium (2):
  - UZ Gent, Ghent
  - Chr de La Citadelle, Liège
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Italy (6):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Policlinico Agostino Gemelli, Rome, Lazio
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Fondazione IRCCS Istituto Neurologico ?Carlo Besta?, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda, Milan, Lombardy
  - Ospedali Riuniti Torrette di Ancona, Ancona, The Marches
- Japan (3):
  - Kobe University Hospital, Hyōgo
  - Kagoshima University Hospital, Kagoshima
  - National Center for Global Health and Medicine, Tokyo
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
- Portugal (2):
  - CHULC, E.P.E. - Hospital Dona Estefania, Lisbon
  - Hospital de Santa Maria, Lisbon
- Spain (4):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario la Fe, Valencia
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Great Ormond Street Hospital For Children, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing